CLINICAL TRIAL: NCT02810249
Title: Factors Affecting the Likely Use of PrEP for African American Young Men Who Have Sex With Men
Brief Title: Likely Use of PrEP for African American YMSM
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00070892
Record Dates: First submitted 2016-05-25; First posted 2016-06-22 (Estimated); Last update posted 2017-04-14 (Actual); Status verified 2017-04

CONDITIONS: HIV
Keywords: African American YMSM; PrEP; HIV Pre-Exposure Prophylaxis; Common Sense Model; Healthcare; HIV Prevention

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- African American YMSM
  Interventions: Other: No intervention used

INTERVENTIONS:
Other: No intervention used

SUMMARY:
HIV Pre-Exposure Prophylaxis (PrEP), in the form of the anti-retroviral pill Truvada©, has been approved by the FDA as a method for reducing HIV transmission rates in the population, particularly young men who have sex with men (YMSM). This study will use a qualitative design to interview 20-30, HIV-negative, 16-24 year old African American YMSM to: 1) identify and understand African American YMSM's, aged 16-24, cognitive and emotional processes in response to using PrEP to reduce their risk for HIV and 2) identify what factors (sociocultural, individual, experiences in health care, socioeconomic) influence African American YMSM's likely use of PrEP as a coping strategy for HIV prevention. Demographic information will be collected and analyzed using Statistical Analysis Software version 9.3. Individual interviews will be audio recorded and transcribed by a vetted transcription service for analysis. This is minimal risk to participants.

DETAILED DESCRIPTION:
This study will use an exploratory, naturalistic qualitative design where participants will be interviewed to collect data on their emotional and cognitive processes (illness representation) in response to the threat of a potential HIV infection, and what factors (social, cultural, individual characteristics, and experiences in health care) influence their likely use of PrEP. The sample for this study will include 20 to 30 African American YMSM, aged 16-24, residing in Durham, Wake, and Orange counties of North Carolina.

The in-depth interview guide and the 26-item descriptive survey PrEP Knowledge, Sexual History, and Demographic Instrument were developed for this study using a combination of the concepts from the adapted Common Sense Model of Illness Representation (CSM) and questions adapted from the Adolescent Trial Network's (ATN) 082 study's questionnaire. Participants will be asked questions relating to African American YMSM's likely use of HIV Pre-Exposure Prophylaxis (PrEP) as an HIV risk-reduction strategy. Once informed consent is obtained, the interview will commence and study participants will be individually interviewed to discuss what factors influence their likely use of PrEP. Each participant will complete the descriptive survey and the one-on-one interview.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 16-24
* self-identify as African-American, Black, or mixed race including African American or Black
* have been assigned male sex at birth
* self-identify as gay, bisexual, or queer, or self-identify as a heterosexual male who has had a past voluntary sexual experience with another man or currently has sexual desires for men
* report being uninfected with HIV
* be mentally capable of providing informed consent
* be able to speak and read English
* not currently using PrEP for HIV.

Exclusion Criteria:

* HIV-infected men are excluded because this study is focused on the prevention of HIV transmission
* Men who were not assigned male sex at birth are excluded from this study, because transgender men face very different and distinct issues with access to care compared to YMSM
* Men who are currently using PrEP are excluded from this study because this study is exploring the barriers and facilitators to use of PrEP in African American YMSM aged 16-24. Men who are currently using PrEP may have a different illness representation compared to men who are not using PrEP.

Ages: 16 Years to 24 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 20 to 30 African American young men who have sex with men, aged 16-24
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2016-12-29 (Actual); Study Completion 2016-12-29 (Actual)

PRIMARY OUTCOMES:
Factors that influence African American YMSM's likely use of PrEP | During patient interview, approximately 1.5 hours
Cognitive processes in response to using PrEP to reduce risk for HIV | During patient interview, approximately 1.5 hours
Emotional processes in response to using PrEP to reduce risk for HIV | During patient interview, approximately 1.5 hours

IPD SHARING:
Plan to Share IPD: No